CLINICAL TRIAL: NCT07284667
Title: A Double-Blind, Placebo-Controlled, Parallel Group, Efficacy and Safety Study of ACP-211 Monotherapy in Adults With Major Depressive Disorder and Inadequate Response to Antidepressant Treatment
Brief Title: ACP-211 Monotherapy for Major Depressive Disorder With Inadequate Antidepressant Response
Acronym: NORLIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-211-002
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD); Depressive Disorder, Treatment-Resistant
Keywords: Major Depressive Disorder (MDD); Depressive Disorder, Treatment-Resistant; Antidepressive Agents; Randomized Controlled Trial; Double-Blind Method; Clinical Trial, Phase II; Psychiatric Status Rating Scales; Ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ACP-211 600 mg (Experimental): ACP-211 600 mg, administered orally twice weekly
  Interventions: Drug: ACP-211
- ACP-211 300 mg (Experimental): ACP-211 300 mg, administered orally twice weekly
  Interventions: Drug: ACP-211
- Placebo (Placebo Comparator): Matching placebo, administered orally twice weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-211 — ACP-211 monotherapy
  Arms: ACP-211 300 mg; ACP-211 600 mg
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if ACP-211 can help treat adults with major depressive disorder (MDD) who have not improved with antidepressant therapy (ADT), including those with treatment resistant depression (TRD).

The main questions the study aims to answer are:

* Does ACP-211 work better than a placebo (a look-alike capsule with no medicine) to reduce symptoms of depression?
* What adverse events do participants have when taking ACP-211?

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 and ≤65 years of age
* Provides written informed consent
* Clinical diagnosis of MDD
* History of inadequate response to at least two antidepressants, with at least one inadequate response documented during the current episode
* Currently treated with an approved antidepressant at a stable dose prior to Screening
* MADRS total score ≥28, CGI-S score ≥4 , and QIDS-SR16 score ≥16 at Screening and Baseline
* Females of childbearing potential must have a negative pregnancy test and agree to use acceptable contraception; males must agree to use barrier protection and refrain from sperm donation

Exclusion Criteria:

* Current diagnosis of certain personality disorders or persistent depressive disorder
* Recent substance use disorders, excluding caffeine or nicotine
* Active suicidal risk or recent suicidal attempt
* History of schizophrenia, psychotic disorders, bipolar disorder, or MDD with psychotic features
* Current treatment requirement for PTSD, acute stress disorder, panic disorder, or OCD
* History of neuroleptic malignant syndrome, serotonin syndrome, or epilepsy (except single febrile seizure in infancy)
* Documented non-response to ADT, including ketamine or esketamine
* Allergy or sensitivity to ketamine or esketamine
* Significant cardiovascular disease
* Positive history of hepatitis B, hepatitis C, or HIV infection
* Unstable diabetes or uncontrolled medical conditions
* Positive urine drug test for an illicit drug or cannabis
* Received neuromodulation therapies (ECT,TMS, VNS, DBS) in the current depressive episode
* Recent initiation or change in psychotherapy Additional inclusion/exclusion criteria apply. Participants will be evaluated at Screening to ensure that all criteria for study participation are met.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at Day 28 | Baseline and Day 28
  The MADRS is a clinician-rated tool that assesses the severity of depressive symptoms. It consists of 10 items, each scored from 0 (no symptoms) to 6 (severe symptoms), resulting in a total score range of 0 to 60. Higher scores indicate greater depression severity.

SECONDARY OUTCOMES:
Change from Baseline in the MADRS total score postdose at 24 hours (Day 2) | Baseline and Day 2

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Inland Psychiatric Medical Group, Chino, California
  - Mountain View Clinical Research, Denver, Colorado
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - IPTB Clinical Research, Tampa, Florida
  - CenExel Hassman Research Institute, LLC, Marlton, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Dynamed Clinical Research LP d/b/a DM Clinical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No